CLINICAL TRIAL: NCT05174169
Title: Colon Adjuvant Chemotherapy Based on Evaluation of Residual Disease
Acronym: CIRCULATE-US
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: Natera, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GI008; U10CA180868 (NIH); NRG-GI008 (Other: NRG Oncology); NCI-2021-08397 (Other: NCI)
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Stage III Colon Cancer
Keywords: ctDNA positive; ctDNA negative; Adjuvant Chemotherapy; Natera; Signatera; mFOLFOX6; Stage III; CAPOX; mFOLFIRINOX; Oxaliplatin; 5-Fluorouracil (5-FU); Capecitabine; Leucovorin; Irinotecan; Stage II
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Cohort A - Arm 1 (ctDNA-ve) (Active Comparator): Oxaliplatin 85 mg/m2 IV + Leucovorin 400mg/m2 IV + 5-Fluorouracil (5-FU) 400mg/m2 bolus + 5-Fluorouracil (5-FU) 2400mg/m2 IV continuous infusion over 46-48 hours (total dose) Day1 every 2 weeks for 6-12 cycles
  OR
  Oxaliplatin 130 mg/m2 IV Day 1 every 3 weeks + Capecitabine 1000 mg/m2 BID by mouth days 1-14 every 3 weeks for 4 cycles
  Interventions: Device: Signatera test; Drug: mFOLFOX6 3-6 month; Drug: CAPOX 3 month
- Cohort A - Arm 2 (ctDNA-ve) (Experimental): Serial ctDNA monitoring no treatment
  Interventions: Device: Signatera test
- Cohort B - Arm 3 (ctDNA+ve) (Active Comparator): Oxaliplatin 85 mg/m2 IV + Leucovorin 400mg/m2 IV + 5-Fluorouracil (5-FU) 400mg/m2 bolus + 5-Fluorouracil (5-FU) 2400mg/m2 IV continuous infusion over 46-48 hours (total dose) Day1 every 2 weeks for 12 cycles
  OR
  Oxaliplatin 130 mg/m2 IV Day 1 every 3 weeks + Capecitabine 1000 mg/m2 BID by mouth days 1-14 every 3 weeks for 8 cycles
  Interventions: Device: Signatera test; Drug: mFOLFOX6 6 month; Drug: CAPOX 6 month
- Cohort B - Arm 4 (ctDNA+ve) (Experimental): Oxaliplatin 85 mg/m2 IV + Leucovorin 400mg/m2 IV + Irinotecan 150 mg/m2 IV continuous infusion (30-90 minutes) + 5-Fluorouracil (5-FU) 2400mg/m2 IV continuous infusion over 46-48 hours (total dose) Day1 every 2 weeks for 12 cycles
  Interventions: Device: Signatera test; Drug: mFOLFIRINOX

INTERVENTIONS:
Device: Signatera test — Central ctDNA testing for all patients
Drug: mFOLFOX6 3-6 month — Oxaliplatin 85 mg/m2 IV + Leucovorin 400mg/m2 IV + 5-Fluorouracil (5-FU) 400mg/m2 bolus + 5-Fluorouracil (5-FU) 2400mg/m2 IV continuous infusion over 46-48 hours (total dose) Day1 every 2 weeks for 6-12 cycles
  Arms: Cohort A - Arm 1 (ctDNA-ve)
Drug: CAPOX 3 month — Oxaliplatin 130 mg/m2 IV Day 1 every 3 weeks + Capecitabine 1000 mg/m2 BID by mouth days 1-14 every 3 weeks for 4 cycles
  Arms: Cohort A - Arm 1 (ctDNA-ve)
Drug: mFOLFIRINOX — Oxaliplatin 85 mg/m2 IV + Leucovorin 400mg/m2 IV + Irinotecan 150 mg/m2 IV continuous infusion (30-90 minutes) + 5-Fluorouracil (5-FU) 2400mg/m2 IV continuous infusion over 46-48 hours (total dose) Day1 every 2 weeks for 12 cycles
  Arms: Cohort B - Arm 4 (ctDNA+ve)
Drug: mFOLFOX6 6 month — Oxaliplatin 85 mg/m2 IV + Leucovorin 400mg/m2 IV + 5-Fluorouracil (5-FU) 400mg/m2 bolus + 5-Fluorouracil (5-FU) 2400mg/m2 IV continuous infusion over 46-48 hours (total dose) Day1 every 2 weeks for 12 cycles
  Arms: Cohort B - Arm 3 (ctDNA+ve)
Drug: CAPOX 6 month — Oxaliplatin 130 mg/m2 IV Day 1 every 3 weeks + Capecitabine 1000 mg/m2 BID by mouth days 1-14 every 3 weeks for 8 cycles
  Arms: Cohort B - Arm 3 (ctDNA+ve)

SUMMARY:
This Phase II/III trial will evaluate the what kind of chemotherapy to recommend to patients based on the presence or absences of circulating tumor DNA (ctDNA) after surgery for colon cancer.

DETAILED DESCRIPTION:
Currently, there are no biomarkers validated prospectively in randomized studies for resected colon cancer to determine need for adjuvant chemotherapy. However, circulating tumor DNA (ctDNA) shed into the bloodstream represents a highly specific and sensitive approach (especially with serial monitoring) for identifying microscopic or residual tumor cells in colon cancer patients and may outperform traditional clinical and pathological features in prognosticating risk for recurrence. Colon cancer patients who do not have detectable ctDNA (ctDNA-) are at a much lower risk of recurrence and may not need adjuvant chemotherapy. Furthermore, for colon cancer pts with detectable ctDNA (ctDNA+) who are at a very high risk of recurrence, the optimal adjuvant chemotherapy regimen has not been established. We hypothesize that for pts whose colon cancer has been resected, ctDNA status may be used to risk stratify for making decisions about adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

The patient must have an ECOG performance status of 0 or 1.

Patients must have histologically/pathologically confirmed Stage IIB, IIC, or Stage III colon adenocarcinoma with R0 resection according to AJCC 8th edition criteria.

No radiographic evidence of overt metastatic disease within 45 days prior to Step 1/Study entry (CT with IV contrast or MRI imaging is acceptable and must include chest, abdomen, and pelvis).

The distal extent of the tumor must be greater than or equal to 12 cm from the anal verge on colonoscopy or above the peritoneal reflection as documented during surgery or on pathology specimen (i.e., excluding rectal adenocarcinomas warranting treatment with chemoradiation).

The patient must have had an en bloc complete gross resection of tumor (curative resection). Patients who have had a two-stage surgical procedure, to first provide a decompressive colostomy and then in a later procedure to have the definitive surgical resection, are eligible.

The resected tumor specimen and a blood specimen from patients with Stage IIB, IIC, or Stage III colon cancer must have central testing for ctDNA using the Signatera™ assay by Natera (after Step 1/Study entry and before Step2/Randomization). Patient must have sufficient tissue to meet protocol requirements. This blood specimen for the Signatera assay must be collected after surgery (and recommended at least 14 days post surgery).

Tumor must be documented as microsatellite stable or have intact mismatch repair proteins through CLIA-approved laboratory testing. Patients whose tumors are MSI-H or dMMR are excluded.

The treating investigator must deem the patient a candidate for all potential agents used in this trial (5FU, LV, oxaliplatin and irinotecan).

The interval between surgery (post-operative Day 7) and Step 1/Study entry must be no more than 60 days. NOTE: Step 1/Study Entry may occur as early as post operative Day 7, but it cannot occur beyond 60 days from the actual date of the patient's surgery.

Availability and provision of adequate surgical tumor tissue for molecular diagnostics and confirmatory profiling.

Adequate hematologic function within 28 days before Step 1/Study entry defined as follows:

* Absolute neutrophil count (ANC) must be greater than or equal to 1500/mm3;
* Participants with benign ethnic neutropenia (BEN): ANC less than 1300 mm3 are eligible.
* BEN (also known as constitutional neutropenia) is an inherited cause of mild or moderate neutropenia that is not associated with any increased risk for infections or other clinical manifestations. BEN is referred to as ethnic neutropenia because of its increased prevalence in people of African descent and other specific ethnic groups.
* Platelet count must be greater than or equal to 100,000/mm3; and
* Hemoglobin must be greater than or equal to 9 g/dL.

Adequate hepatic function within 28 days before Step 1/Study entry defined as follows:

* total bilirubin must be less than or equal to ULN (upper limit of normal) for the lab and
* alkaline phosphatase must be less than 2.5 x ULN for the lab; and
* AST and ALT must be less than 2.5 x ULN for the lab.

Adequate renal function within 28 days before Step 1/Study entry defined as serum creatinine less than or equal to 1.5 x ULN for the lab or measured or calculated creatinine clearance greater than or equal to 50 mL/min using the Cockroft-Gault formula for patients with creatinine levels greater than 1.5 x ULN for the lab.

For Women Creatinine Clearance (mL/min) = (140 - age) x weight (kg) x 0.85 72 x serum creatinine (mg/dL) For Men Creatinine Clearance (mL/min) = (140 - age) x weight (kg) 72 x serum creatinine (mg/dL) NOTE: Adjusted body weight (AdjBW) should be used for patients that have BMI greater than or equal to 28 (less than or equal to 30% above IBW).

HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.

Pregnancy test (urine or serum according to institutional standard) done within 14 days before Step 1/Study entry must be negative (for women of childbearing potential only).

Patients receiving a coumarin-derivative anticoagulant must agree to weekly monitoring of INR if they are randomized to Arm 1 or Arm 3 and receive capecitabine.

Eligibility Criteria for Cohort A Arm-2 patients on Second Randomization

Patient must have developed a ctDNA +ve assay during serial monitoring.

Patient's willingness to be re-randomized affirmed.

The patient must continue to have an ECOG performance status of 0 or 1.

No radiographic evidence of overt metastatic disease.

Pregnancy test (urine or serum according to institutional standard) done within 14 days before second randomization must be negative (for women of childbearing potential only).

Adequate hematologic function within 28 days before second randomization defined as follows:

* Absolute neutrophil count (ANC) must be greater than or equal to 1500/mm3;
* Participants with benign ethnic neutropenia (BEN): ANC less than 1300 mm3 are eligible.
* BEN (also known as constitutional neutropenia) is an inherited cause of mild or moderate neutropenia that is not associated with any increased risk for infections or other clinical manifestations. BEN is referred to as ethnic neutropenia because of its increased prevalence in people of African descent and other specific ethnic groups.
* Platelet count must be greater than or equal to 100,000/mm3; and
* Hemoglobin must be greater than or equal to 9 g/dL.

Adequate hepatic function within 28 days before second randomization defined as follows:

* total bilirubin must be less than or equal to ULN (upper limit of normal) for the lab and
* alkaline phosphatase must be less than 2.5 x ULN for the lab; and
* AST and ALT must be less than 2.5 x ULN for the lab.

Adequate renal function within 28 days before second randomization defined as serum creatinine less than or equal to 1.5 x ULN for the lab or measured or calculated creatinine clearance greater than or equal to 50 mL/min using the Cockroft-Gault formula for patients with creatinine levels greater than 1.5 x ULN for the lab.

For Women Creatinine Clearance (mL/min) = (140 - age) x weight (kg) x 0.85 72 x serum creatinine (mg/dL) For Men Creatinine Clearance (mL/min) = (140 - age) x weight (kg) 72 x serum creatinine (mg/dL)

Exclusion Criteria:

Colon cancer histology other than adenocarcinoma (i.e., neuroendocrine carcinoma, sarcoma, lymphoma, squamous cell carcinoma, etc.).

Pathologic, clinical, or radiologic overt evidence of metastatic disease. This includes isolated, distant, or non-contiguous intra-abdominal metastases, even if resected.

Tumor-related bowel perforation.

History of prior invasive colon malignancy, regardless of disease-free interval.

History of bone marrow or solid organ transplantation (regardless of current immunosuppressive therapy needs). Bone grafts, skin grafts, corneal transplants and organ/tissue donation are not exclusionary.

Any prior systemic chemotherapy, targeted therapy, or immunotherapy; or radiation therapy administered as treatment for colorectal cancer (e.g., primary colon adenocarcinomas for which treatment with neoadjuvant chemotherapy and/or radiation is warranted are not permitted). EXCEPTION: one cycle of chemotherapy (regimen per treating physicians' discretion - 5-FU or capecitabine with or without oxaliplatin) is allowed but not required after consent. The optional cycle of chemotherapy should be started greater than or equal to 4 weeks from surgery and while awaiting Step 2 randomization.

Other invasive malignancy within 5 years before Step 1/Study entry. Exceptions are colonic polyps, non-melanoma skin cancer or any carcinoma-in-situ.

Synchronous primary rectal and/ or colon cancers.

Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.

Sensory or motor neuropathy greater than or equal to grade 2, according to CTCAE v5.0.

Blood transfusion within two weeks before collection of blood for central ctDNA testing.

Active seizure disorder uncontrolled by medication.

Active or chronic infection requiring systemic therapy.

Known homozygous DPD (dihydropyrimidine dehydrogenase) deficiency.

Patients known to have Gilbert's Syndrome or homozygosity for UGT1A1*28 polymorphism.

Pregnancy or lactation at the time of Step 1/Study entry.

Co-morbid illnesses or other concurrent disease that would make the patient inappropriate for entry into this study (i.e., unable to tolerate 6 months of combination chemotherapy or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens or prevent required follow-up).

Ineligibility Criteria for Cohort A Arm-2 patients on Second Randomization

Pregnancy or lactation at the time of randomization.

No longer a candidate for systemic chemotherapy (FOLFOX, CAPOX, and mFOLFIRINOX) in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1912 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2029-03-10 (Estimated); Study Completion 2030-03-10 (Estimated)

PRIMARY OUTCOMES:
ctDNA positive status (TTPos) | Time from randomization to the first TTPos event, a maximum of 3 years
  TTPos is defined as time from randomization until ctDNA positive event: TTPos events are first ctDNA positive result after randomization for the immediate adjuvant chemo arm (Arm 1), 2nd ctDNA positive result after randomization for the delayed adjuvant chemo (Arm 2) and recurrence without a positive ctDNA result for both arms.
Disease-Free Survival (DFS) | Time from randomization to disease-free survival event, a maximum of 5 years]
  Time from randomization to first disease-free survival event (recurrence, second primary colorectal cancer or death from any cause).

SECONDARY OUTCOMES:
Baseline post-surgery ctDNA positivity rate | At time of randomization
  percentage of patients with ctDNA positive results post-surgery at study entry.
Overall Survival (OS) | Time from randomization to death, a maximum of 5 years.
  Time from randomization to death of any cause.
Recurrence | Time from randomization to disease recurrence, a maximum of 5 years
  Time from randomization to disease recurrence.
Compliance with adjuvant chemotherapy | from randomization to the last cycle of chemotherapy, a maximum of 6 months.
  number of cycles of chemotherapy received.

CONTACTS AND LOCATIONS:
Locations (1034):
- United States (999):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Marshall Cancer Center, Cameron Park, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Epic Care-Dublin, Dublin, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Washington Hospital, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - UCI Health Laguna Hills, Laguna Hills, California
  - City of Hope Antelope Valley, Lancaster, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Loma Linda Healthcare System, Loma Linda, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Mills Health Center, San Mateo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Santa Cruz Radiation Oncology Medical Group, Santa Cruz, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - City of Hope South Bay, Torrance, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - BASS Medical Group - Lennon, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Intermountain Health Platte Valley Hospital, Brighton, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - UCHealth - Cherry Creek, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Dillon Health Center/Shaw Cancer Center, Dillon, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Lutheran Hospital - Cancer Centers of Colorado, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - UCHealth Lone Tree Health Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - AdventHealth Celebration, Celebration, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - Orlando Health Cancer Institute - Lake Mary, Lake Mary, Florida
  - The Watson Clinic, Lakeland, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Tampa General Hospital, Tampa, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Eisenhower Army Medical Center, Fort Eisenhower, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Piedmont Newnan Hospital, Newnan, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Piedmont Henry Hospital, Stockbridge, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - UChicago Medicine AdventHealth Cancer Institute Hinsdale, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Rush MD Anderson Cancer Center at Rush Lisle, Lisle, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center, Moline, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Rush MD Anderson Cancer Center at Rush Oak Park, Oak Park, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Reid Health, Richmond, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Baptist Health Hamburg, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Norton Audubon Hospital and Medical Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - UM Upper Chesapeake Hematology and Oncology - Aberdeen, Aberdeen, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - FMH James M Stockman Cancer Institute, Frederick, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Kaiser Permanente Lutherville - Timonium Medical Center, Lutherville, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Dana-Farber Cancer Institute at Foxborough, Foxborough, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Dana Farber-Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - The Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Summit Medical Group, Berkeley Heights, New Jersey
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - Jefferson Cherry Hill Hospital, Cherry Hill, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Trinitas Hospital and Comprehensive Cancer Center - Williamson Street Campus, Elizabeth, New Jersey
  - Summit Health - Florham Park Campus, Florham Park, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health Cancer Institute at Huntington, Greenlawn, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Queens Cancer Center, Rego Park, New York
  - Rochester General Hospital, Rochester, New York
  - Unity Park Ridge Campus, Rochester, New York
  - University of Rochester, Rochester, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Staten Island University Hospital, Staten Island, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Mount Sinai South Nassau, Valley Stream, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Duke Cancer Center Cary, Cary, North Carolina
  - UNC Health Cancer Care Cary, Cary, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - UNC Health Cancer Care Garner, Garner, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - UNC Health Cancer Care Raleigh, Raleigh, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - UNC Health Cancer Care Wakefield, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Mount Carmel New Albany Surgical Hospital, New Albany, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Mercy Health Sylvania Radiation Oncology Center, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Camp Hill, Camp Hill, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant - Cranberry, Cranberry Township, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Jefferson Methodist Hospital, Philadelphia, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Avera Cancer Institute - Mitchell, Mitchell, South Dakota
  - Avera Cancer Institute at Pierre, Pierre, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Avera Cancer Institute at Yankton, Yankton, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - The West Clinic - Wolf River, Germantown, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Thompson Oncology Group-Oak Ridge, Oak Ridge, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - University of Texas at Austin, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - STCC at DHR Health Institute for Research and Development, Edinburg, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - Cancer Specialists of Tidewater Limited, Chesapeake, Virginia
  - Peninsula Cancer Institute-Gloucester, Gloucester, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Cancer Specialists of Tidewater-Suffolk, Suffolk, Virginia
  - Peninsula Cancer Institute-Cancer Specialists of Tidewater, Virginia Beach, Virginia
  - Peninsula Cancer Institute-Williamsburg, Williamsburg, Virginia
  - Kaiser Permanente-Caton Hill Medical Center, Woodbridge, Virginia
  - FHCC Overlake, Bellevue, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Valley Medical Center, Renton, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - Marshfield Medical Center - Neillsville, Neillsville, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- Canada (30):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - BCCA-Cancer Centre for the North, Prince George, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA-Vancouver Island Cancer Centre, Victoria, British Columbia
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Waterloo Regional Health Network, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Niagara Health System-Saint Catharines General, Saint Catharines, Ontario
  - North York General Hospital, Toronto, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - Hotel-Dieu De Levis, Lévis, Quebec
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Puerto Rico (5):
  - Pan American Center for Oncology Trials LLC - Cayey, Cayey
  - Pan American Center for Oncology Trials LLC - Dorado, Dorado
  - Pan American Center for Oncology Trials LLC - Mayag��ez, San Juan
  - Pan American Center for Oncology Trials LLC, San Juan
  - Pan American Center for Oncology Trials LLC - Ciudadela, San Juan